CLINICAL TRIAL: NCT05589298
Title: Questionnaire on Self-reported Experience of Koebner and Deep-Koebner Phenomenon in Patients With Psoriasis and Psoriatic Arthritis.
Brief Title: The Study of Koebner in Patients With Psoriasis and Psoriatic Arthritis
Acronym: PSODEEP1
Status: Completed | Type: Observational
Sponsor: Skane University Hospital (Other)
Collaborators: University of Chile (Other); University of Copenhagen (Other); Karolinska Institutet (Other); Lund University (Other)
Responsible Party: Principal Investigator, Albert Duvetorp, Principal Investigator, Head of Psoriasis outpatient clinic Malmö, MD PhD, Skane University Hospital
Other Study IDs: PSODEEP1
Record Dates: First submitted 2022-10-15; First posted 2022-10-21 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Psoriasis; Psoriasis; Arthritis (Etiology); Koebner Phenomenon
Keywords: Koebner; Deep-Koebner; Psoriasis; Arthritis
MeSH Terms: conditions — Psoriasis; Arthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- PSODEEP1 Sweden: Patients with self reported MD given diagnosis of psoriasis and/or psoriatic arthritis in Sweden.
- PSODEEP1 Denmark: Patients with self reported MD given diagnosis of psoriasis and/or psoriatic arthritis in Denmark.
- PSODEEP1 Chile: Patients with self reported MD given diagnosis of psoriasis and/or psoriatic arthritis in Chile.
- PSODEEP1 Netherlands: Patients with self reported MD given diagnosis of psoriasis and/or psoriatic arthritis in the Netherlands.

SUMMARY:
PSODEEP 1 is a descriptive digital interview study where we intend to include at least 900 individuals. Individuals with known psoriasis or known psoriatic arthritis will access the digital interview via a QR code distributed via their rheumatology or dermatology department using their smartphones. Data on answers results are stored digitally and can be accessed parallel to recruitment. Questions focus on following fields (all self reported): background information (age/sex), disease duration, disease course/fluctuation, disease diagnosis as given by MD, disease treatment, disease severity, disease classification, disease triggers, screening of psoriatic arthritis (questions derived from PEST questionnaire), Koebner occurence, variability in Koebner over time, deep-Koebner occurence and variability in Deep-Koebner over time.

DETAILED DESCRIPTION:
PSODEEP1 is a descriptive digital interview study. Questions on self reported experience of following fields will be stated: background information, disease duration, disease course/fluctuation, disease diagnosis as given by MD, disease treatment, disease severity, disease classification, disease triggers, screening of psoriatic arthritis (questions derived from PEST questionnaire), Koebner occurence, variability in Koebner over time, deep-Koebner occurence and variability in Deep-Koebner over time.

Questions will be distributed using REDCap (REsearch Electronic Data CAPture) platform provided by Lunds university, University of Santiago and Copenhagen University (www.project-redcap.org). Patients with known psoriasis or psoriatic arthritis will reach the questionnaire using a QR-code on patient's information sheet distributed in clinical settings. In Sweden, patients will be recruited at dermatology and rheumatology outpatient clinics in Malmö, Lund, Göteborg, Örebro, Stockholm (Skåne University Hospital, Karolinska Hospital, Sahlgrenska Hospital, Ryhov Hospital, Örebro, Hospital). In Chile patients will be recruited at Hospital Clínico Universidad de Chile and CIEC-PMR Centro Internacional de Estudios Clínicos - Probity Medical Research. In Denmark, patients will be recruited at Gentofte Hospital and through Leo foundation skin immunology research center (Copenhagen University) and the Parker Institute.

Study inclusion criteria: Physician diagnosed psoriasis, psoriatic arthritis or both. Age of 18 years or older. Ability to comprehend instructions and read the Swedish, Spanish or Danish language (according to country). Having a smartphone with which one can access the study questions using a QR code. Study exclusion criteria: Having participated in the study already. Not having a mobile telephone number (used to identify duplicate answers).

ELIGIBILITY:
Inclusion Criteria:

* MD diagnosis of psoriasis and/or psoriasis arthritis
* Age over 18 years
* Ability to read and understand written questions
* Having/ability to use smartphone
* Given consent

Exclusion Criteria:

- Having participated previously

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with psoriasis and/or psoriatic arthritis
Sampling Method: Non-Probability Sample
Enrollment: 3064 (Actual)
Dates: Start 2022-10-19 (Actual); Primary Completion 2024-02-14 (Actual); Study Completion 2024-02-14 (Actual)

PRIMARY OUTCOMES:
Koebner | Through study completion, estimated to 12 months.
  Occurence of Self-Reported Koebner phenomena. Self-reported in multiple choice questionnaire "Has your skin psoriasis ever developed at the site of a skin injury, such as a scrape or a burn?" YES/NO/DO NOT KNOW. Ordinal data.
Trauma induced Deep-Koebner | Through study completion, estimated to 12 months.
  Occurence of Self-Reported trauma induced Deep-Koebner phenomena in patients with with psoriasis arthritis. Questionnaire, self-reported, multiple choice "Have you ever developed psoriatic arthritis in a joint after injury, e.g. after a fall or sprain? " YES/NO/DO NOT KNOW. Ordinal data.

SECONDARY OUTCOMES:
Variation in Koebner | Through study completion, estimated to 12 months.
  Variation of self-reported Koebner over time. In patients with self-reported Koebner a following multiple choice question will assess if Koebner is a constant phenomenon or whether it is associated with periods of high psoriasis disease activity. Multiple choice answers, self-reported, collected in questionnaire. Ordinal data.
Variation in Trauma induced Deep-Koebner | Through study completion, estimated to 12 months.
  Variation of self-reported Trauma induced Deep-Koebner over time. In patients with self-reported trauma induced Deep-Koebner a following multiple choice question will assess if Deep-Koebner is a constant phenomenon or whether it is associated with periods of high psoriasis disease activity. Answer is multiple choice, self-reported. Ordinal data.

OTHER OUTCOMES:
Worsening of psoriasis due to scratching | Through study completion, estimated to 12 months.
  Self-reported, multiple choice answer in questionnaire "Does your skin psoriasis worsen due to scraping or scratching (e.g. secondary to itch)?" YES/NO/DO NOT KNOW. Ordinal data.
Variation in worsening of psoriasis due to scratching over time | Through study completion, estimated to 12 months.
  Follow up question to participants that report worsening due to scratching. Multiple choice question in order to assess if this experience is constant or related to overall disease activity. Ordinal data.
Presence of symptoms that could imply presence of psoriatic arthritis. | Through study completion, estimated to 12 months.
  Multiple choice questions in digital questionnaire assessing self-reported presence of dactylitis, nail-pitting, tendinitis and arthritis. Output is ordinal data.

CONTACTS AND LOCATIONS:
Overall Officials: Albert Duvetorp, MD PhD, Principal Investigator — Lunds University, Copenhagen University
Locations (1):
- Hudkliniken Skånes Universitetssjukhus, Malmo, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
Data can be shared upon reasonable request if the correct legal arrangements can be set up (according to GDPR and data protection laws etc).

REFERENCES:
- [Background] Weiss G, Shemer A, Trau H. The Koebner phenomenon: review of the literature. J Eur Acad Dermatol Venereol. 2002 May;16(3):241-8. doi: 10.1046/j.1473-2165.2002.00406.x. PMID 12195563
- [Background] Soltani-Arabshahi R, Wong B, Feng BJ, Goldgar DE, Duffin KC, Krueger GG. Obesity in early adulthood as a risk factor for psoriatic arthritis. Arch Dermatol. 2010 Jul;146(7):721-6. doi: 10.1001/archdermatol.2010.141. PMID 20644032
- [Background] Pattison E, Harrison BJ, Griffiths CE, Silman AJ, Bruce IN. Environmental risk factors for the development of psoriatic arthritis: results from a case-control study. Ann Rheum Dis. 2008 May;67(5):672-6. doi: 10.1136/ard.2007.073932. Epub 2007 Sep 6. PMID 17823200